CLINICAL TRIAL: NCT04018430
Title: Impact d'Une Surcharge Glycemique Sur le Taux HbA1c
Brief Title: Impact of Oral Glucose Tolerance Test on Extent of Hemoglobin Glycation
Acronym: HbA1c
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Urs E. Nydegger (Industry)
Collaborators: Labormedizinisches Zentrum Dr. Risch (Industry)
Responsible Party: Sponsor-Investigator, Urs E. Nydegger, Head Hematology Senior Consultant, Labormedizinisches Zentrum Dr. Risch
Organization: Labormedizinisches Zentrum Dr. Risch (Industry)
Other Study IDs: Lmzrisch
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Blood Glucose, High; Oral Hypoglycaemic Overdose
Keywords: glucose, insulin, HbA1c
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Days
Biospecimen Retention: Samples Without DNA — venous blood samples processed to yield 4 ml of blood plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The glycation extent of human hemoglobin is under control of the Maillard reaction, a chemical interaction between an amino acide and a reducing sugar. About 5% ( 31.1 mmol/mol) of hemoglobin molecules secluded in a red blood cell are glycated; excessive values > 6.5% point to prediabetes or overt diabetes mellitus. To ascertain the diagnosis doctors prescribe oral glucose tolerance upon which glucose concentrations in blood increase - how much HbA1c reacts under these circumstances is ill known.

DETAILED DESCRIPTION:
Medical laboratory assays for delineation of impaired glucose metabolism and overt diabetes mellitus, beyond measurement of (fasting) blood serum or plasma glucose levels, include extent of hemoglobin A1c glycation, concentration of fructosamines, insulin concentrations to calculate the homeostasis model assessment (HOMA) index and other clinically putative biomarkers of glucose homoeostasis. HbA1c levels form now part of routine elucidation of metabolic disorders and are used for therapy monitoring. Initially used to monitor glucose levels in follow-up care of diabetics it is considered as a track marker of ups and downs of blood glucose concentrations. Its behavior under the 2 h period of oral glucose tolerance tests (OGTT) is ill known - most clinicians believe the glycation extent will not change. Since the dynamics of glycation is temperature dependent,non-febrile patients under OGTT likely keep their glycation extent between time zero and 120 min after glucose charge constant but this has not been investigated and with the sensitive lab assays for HbA1c now in use we postulate a significant increase in glycation. The Patient Registry includes recruited children and adults sick from diabetes, overweight or metabolic syndrome as a whole. Three medical offices will address their patients to the VidyMed lab to perform the OGTT framed by lab assays on venous blood samples

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy subjects or subjects supposedly experiencing a metabolic disease (e.g. prediabetes) Subjects with asked for fasting blood glucose

Exclusion Criteria:

* current steroid use thyroid dysfunction (free-thyroxin levels < 9 or > 19 pmol/L, hsCRP > 10 mg/L hospitalized

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: (i) Those suspected to suffer from the metabolic syndrome including high blood pressure, high blood sugar, excess of body fat and increased cholesterol levels (ii) patients with overt impaired carbohydrate metabolisms, under treatment and tested for follow up
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c concentration upon oral glucose tolerance testing | 48 hours
  HbA1c significantly increases upon oral glucose tolerance testing

CONTACTS AND LOCATIONS:
Overall Officials: Urs Nydegger, MD, Study Chair — Labormedizinisches Zentrum Dr. Risch
Locations (1):
- University of Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
peer reviewed publication in an anglophone scientific journal. No IPD sharing

REFERENCES:
- [Background] Medina Escobar P, Moser M, Risch L, Risch M, Nydegger UE, Stanga Z. Impaired glucose metabolism and type 2 diabetes in apparently healthy senior citizens. Swiss Med Wkly. 2015 Nov 23;145:w14209. doi: 10.4414/smw.2015.14209. eCollection 2015. PMID 26594954
- [Background] Rabbani N, Ashour A, Thornalley PJ. Mass spectrometric determination of early and advanced glycation in biology. Glycoconj J. 2016 Aug;33(4):553-68. doi: 10.1007/s10719-016-9709-8. Epub 2016 Jul 20. PMID 27438287